CLINICAL TRIAL: NCT06687382
Title: A Phase IIa Randomized, Controlled, Open-label Clinical Trial to Assess the Efficacy, Safety, and Tolerability of the Investigational Medicinal Product MBK-01, FSPIM (Full Spectrum & Purified Intestinal Microbiota) Oral Capsules, as Well as to Determine the Optimal Dosage in the Treatment of Patients With Recurrent Diverticulitis (DIREBIOT)
Brief Title: Clinical Trial With MBK-01, Intestinal Microbiota Capsules, for the Treatment of Patients With Recurrent Diverticulitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mikrobiomik Healthcare Company S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIREBIOT; 2023-506224-87-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-31; First posted 2024-11-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Diverticulitis; Diverticulitis of Sigmoid
Keywords: Recurrent Diverticulitis; Diverticular Disease; Acute Diverticulitis; Diverticulosis; Fecal Microbiota Transplantation; Fecal Microbiota Transfer; Intestinal Microbiota
MeSH Terms: conditions — Diverticulitis; Diverticular Diseases; Diverticulum | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MBK-01 with no maintenance dose (Experimental): Participants will receive MBK-01 capsules of intestinal microbiota coming from healthy donors. They will receive an initial dose of 4 capsules the first day, followed by a single daily capsule during 16 days.
  Interventions: Biological: MBK-01
- MBK-01 with maintenance dose (Experimental): Participants will receive MBK-01 capsules of intestinal microbiota coming from healthy donors. They will receive an initial dose of 4 capsules the first day, followed by a single daily capsule during 16 days. 3 months after the ending of the initial dose they will receive a maintenance dose, administered the same as the initial dose.
  Interventions: Biological: MBK-01
- No intervention (No Intervention): Participants will not receive any intervention.

INTERVENTIONS:
Biological: MBK-01 — Initial dose of 4 capsules of MBK-01 (heterologous lyophilized intestinal microbiota coming from healthy donors) orally the first day, followed by a single daily capsule during 16 days. Participants will receive a total dose of 20 capsules of MBK-01.
  Other Names: Fecal Microbiota Transplantation; Intestinal Microbiota Transplantation
  Arms: MBK-01 with no maintenance dose
Biological: MBK-01 — Initial dose of 4 capsules of MBK-01 (heterologous lyophilized intestinal microbiota coming from healthy donors) orally the first day, followed by a single daily capsule for 16 days and a maintenance dose 3 months after the ending of the initial dose. The maintenance dose is administered the same as the initial dose: 4 capsules of MBK-01 orally the first day, followed by a single daily capsule for 16 days. Participants will receive a total dose of 40 capsules of MBK-01.
  Other Names: Fecal Microbiota Transplantation; Intestinal Microbiota Transplantation
  Arms: MBK-01 with maintenance dose

SUMMARY:
Patients with diverticulitis experience a prolonged course of the disease and report a variety of physical, psychological and social symptoms, which highly impacts in their quality of life. Although antibiotic therapy has been the preferred treatment option for acute diverticulitis, it does not control the disease in 40 percent of the patients with complicated diverticulitis and 13 to 23 percent of the patients with non-complicated diverticulitis, which results in chronic and recurrent episodes of diverticulitis. As the episodes repeat, the outpatient conservative treatment has worse success rates and the incidence of complicated diverticulitis with abscess increases up to five times.

Therefore, it is of great importance to establish new treatments in order to avoid the recurrences of the disease. As of today, there is not enough evidence of the efficacy of current treatment options to prevent recurrences in patients with diverticulitis, but recent approaches suggest the modification of intestinal microbiota as a preventive strategy.

Microbial imbalance (dysbiosis) has been proposed as a mechanism involved in the transition from diverticulosis to diverticulitis, inflammation and some of the symptoms of the disease. In this way, fecal microbiota transplantation (FMT) could have an important role in the prevention of new episodes, as it can modify the composition of the intestinal microbiota in a less invasive and more physiological way. Until now the efficacy of FMT in patients with recurrent diverticulitis has not been assessed; however, its benefits and safety have been demonstrated in studies for inflammatory bowel disease (IBD), a pathology with similarities to diverticulitis in its symptoms and underlying inflammation.

The objective of the present clinical trial is to assess the efficacy of MBK-01 (heterologous lyophilized intestinal microbiota oral capsules) in reducing the frequency of episodes in recurrent diverticulitis, its safety and tolerability and to determine the optimal dosing regimen.

DETAILED DESCRIPTION:
This is a phase IIa, randomized, controlled, open-label clinical trial with three treatment arms.

After an initial phase of screening, participants with recurrent diverticulitis will be randomly assigned (1:1:1) to one of the following arms:

* Experimental group with MBK-01 (heterologous lyophilized intestinal microbiota) and no maintenance dose.
* Experimental group with MBK-01 and maintenance dose.
* Control group with no intervention.

Participants assigned to the experimental groups that receive MBK-01 will receive a pre-treatment with antibiotics that consists in the administration of amoxicillin 500 mg (1500 mg/day), fosfomycin 500 mg (3000 mg/day) and metronidazole 250 mg (750 mg/day) for 3 days. After those 3 days, participants will have a washout period of 2 days prior to starting the treatment with MBK-01.

Experimental group with MBK-01 and no maintenance dose will receive an initial dose of 4 oral capsules of MKB-01 in the first day, followed by a daily capsule during the next 16 days. In total, the participant will receive 20 capsules of MBK-01.

Experimental group with MBK-01 and maintenance dose will receive an initial dose of 4 oral capsules of MBK-01 in the first day, followed by a daily capsule during the next 16 days and a maintenance dose 3 months after finishing with the initial dose. The maintenance dose will be administered the same as the initial dose: 4 oral capsules in the first day, followed by a daily capsule during the next 16 days. In total, the participant will receive 40 oral capsules of MBK-01.

Control group with no intervention will not receive any medication oriented to prevent the recurrence of the episodes of diverticulitis.

Regardless of the treatment group to which they have been assigned, all participants will receive the usual rescue antibiotic treatment in the disease when a new episode occurs, and they can also receive the usual support measures they need during the episode (e.g. gastric protection diet or analgesics).

Objectives:

* To assess the efficacy of MBK-01 and its different dosing regimens compared to the control group in reducing the frequency of episodes of acute diverticulitis.
* To assess the safety and tolerability of MBK-01 in its different dosing regimens in patients with diverticulitis.
* To determine the optimal dosing regimen of MBK-01.
* To assess the effect of capsule-based FMT on patient-perceived health outcomes.

Follow up:

In addition to the initial screening visit, participants will attend to a total of 6 follow-up visits for 1 year. After the first follow-up visit, they will attend to the clinic after 1 week, 4 weeks, 16 weeks (3 months for group 2), 6 months and 1 year. During these visits: physical examination, anthropometric measurements, laboratory tests and stool samples will be taken; therapeutic adherence, acute diverticulitis episodes, hospitalizations due to acute diverticulitis and need of surgery due to acute diverticulitis will be evaluated; Gastrointestinal Quality of Life Index (GIQLI) and Short Form-36 (SF-36) questionnaires will be performed and adverse events will be monitored.

Rationale: fecal microbiota transplantation can treat the dysbiosis produced in diverticular disease by restoring the intestinal microbiota, regulating the immune system and improving the intestinal barrier function; the treatment of this dysbiosis could reduce the episodes in recurrent diverticulitis.

Donors: All donors are screened to ensure they meet the strict requirements necessary to maintain the safety of the MBK-01.

Justification:

Diverticulosis and acute diverticulitis are considered multifactorial origin diseases, affected by genetics, diet, microbial imbalance (dysbiosis), acute and chronical inflammation, altered colonic motility and neuromuscular alterations.

Current treatment of diverticular disease includes dietary fiber and pharmacological treatment with broad-spectrum antibiotics, anti-inflammatories and probiotics (alone or in combination). In addition, surgery is contemplated in severe cases.

Although antibiotic therapy has been the preferred treatment option for acute diverticulitis, it does not control the disease in 40 percent of the patients with complicated diverticulitis and 13-23% of the patients with non-complicated diverticulitis, which results in chronic and recurrent episodes of diverticulitis. As the episodes repeat, the outpatient conservative treatment has worse success rates and the incidence of complicated diverticulitis with abscess increases up to five times. Therefore, it is of great importance to establish new treatments in order to avoid the recurrence of the disease.

A preventive treatment regimen for recurrent episodes of diverticulitis has not been established yet. However, some strategies have been suggested, such as: lifestyle changes, high fiber diet, treatment with rifaximin, mesalazine and probiotics, and avoiding NSAIDs.

Microbial imbalance (dysbiosis) has been proposed as a mechanism involved in the transition from diverticulosis to diverticulitis, inflammation and some of the symptoms of the disease. It has been established that dysbiosis can lead to inflammation of the mucosa, neuromuscular dysfunction and a deterioration in the intestinal barrier. Changes in microbiota are associated with other digestive diseases, such as inflammatory bowel disease (IBD), irritable bowel syndrome (IBS) and Clostridioides difficile infections (CDI), which have a similar clinical presentation to diverticulitis.

Fecal microbiota transplantation could have an important role in the prevention of new episodes of diverticulitis, through the regulation of this dysbiosis. The efficacy of FMT for the treatment IBD and CDI has been clinically demonstrated, and there are also clinical trials with probiotics that show an improvement of the symptomatology in diverticular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 18-70 (both included).
* Three or more episodes compatible with a diagnosis of acute diverticulitis of the left or sigmoid colon in the 3 years prior to signing the informed consent. The diagnosis of each episode of diverticulitis must have been made by demonstrating inflammation in the colon compatible with diverticulitis in an imaging test (computed tomography or ultrasound) and presenting at least one of the following analytical or clinical alterations :abdominal pain, vomiting, intestinal obstruction, body temperature over 38ºC, constipation (less than one bowel movement every 3 days), elevated acute-phase reactants (leukocytes higher than 11,000 cells/µL and/or C-reactive protein (CRP) higher than 5mg/dL and/or procalcitonin higher than 0.2), rectal bleeding.
* Not having had any symptomatic episode of acute diverticulitis in the 30 days prior to signing the informed consent.
* In the case of women and men of reproductive age, for safety, those who agree to follow the required contraceptive measure from the signing of the informed consent until the penultimate visit of the follow-up period.
* Patients who have signed the informed consent, either autonomously or through a legal representative.

Exclusion Criteria:

* Patients for who the information on episodes of acute diverticulitis required for inclusion in the study cannot be fully verified.
* Patients with acute diverticulitis in the ascending colon, transverse colon or other locations other than the descending or sigmoid colon.
* Previous colonic resection of any segment of the colon.
* Medical history of colorectal cancer.
* Having taken a mechanical colonic preparation in the 3 months prior to signing the informed consent.
* History of abdominal surgery.
* Allergy or intolerance to any component of the investigational medicinal product or ancillary medicinal products (amoxicillin, clavulanic acid, fosfomycin or metronidazole) used in the trial.
* Prior administration of fecal microbiota transplantation (FMT).
* Systemic antibiotic treatment in the 30 days prior to signing the informed consent.
* Taking a marketed probiotic/prebiotic/symbiotic in the 30 days prior to signing the informed consent.
* Treatment with rifaximin or mesalazine in the 30 days prior to signing the informed consent.
* Presence of hereditary or acquired immunodeficiency.
* Chronic infectious diseases such as hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV).
* Pregnancy or lactation.
* Any other condition that, in the opinion of the investigator, could prevent or hinder compliance with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of new episodes of acute diverticulitis during the trial | Up to 1 year after the start of the treatment
  Diagnosis of the new episode by diagnostic imaging (computed tomography scan or ultrasound) and the presence of at least one of the following symptoms: abdominal pain, vomits, intestinal obstruction, body temperature over 38ºC, constipation, elevated acute-phase reactants leukocytes higher than 11,000 cells/µL and/or C-reactive protein higherthan 5mg/dl and/or procalcitonin higher than 0.2), hematochezia reported by the patient.
Time to first episode of acute diverticulitis | Up to 1 year after the start of the treatment
  Time in weeks from the signing of the informed consent to the first episode of acute diverticulitis.
Time to successive episodes of acute diverticulitis (other than the first episode) | Up to 1 year after the start of the treatment
  Time in weeks from the signing of the informed consent to successive episodes of acute diverticulitis (different from the first episode).
Time between episodes of acute diverticulitis | Up to 1 year after the start of the treatment
  Time in weeks between episodes of acute diverticulitis during the trial.
Number of hospitalizations due to acute diverticulitis in the trial | Up to 1 year after the start of the treatment
  Number of hospitalizations because of acute diverticulitis during the trial.
Number courses of systemic antibiotic treatment used in the trial for the episodes of acute diverticulitis | Up to 1 year after the start of the treatment
  Number of systemic antibiotic treatment cycles used during the trial for the episodes of acute diverticulitis.
Need for surgery for acute diverticulitis during the trial | Up to 1 year after the start of the treatment
  Number of patients that abandon the study because of the need for surgery for acute diverticulitis.
Occurrence of Adverse Events (AES) | Up to 1 year after the start of the treatment
  Frequency of AES.
Occurrence of Serious Adverse Events (SAES) | Up to 1 year after the start of the treatment
  Frequency of SAES.
Occurrence of AES that result in discontinuation of study treatment | Up to 1 year after the start of the treatment
  Frequency of AES that result in discontinuation of study treatment.
Occurrence of AES of special interest (AESI) | Up to 1 year after the start of the treatment
  Frequency of AESI.
Occurrence of diverticulitis-related AES | Up to 1 year after the start of the treatment
  Frequency of diverticulitis-related AES.
Changes in vital signs | Up to 1 year after the start of the treatment
  Frequency of patients with abnormal changes in vital signs (systolic blood pressure, diastolic blood pressure, body temperature and heart rate).
Changes in laboratory values | Up to 1 year after the start of the treatment
  Frequency of patients with abnormal changes in laboratory values (biochemical, hematological and coagulation, lipidic, thyroid, hepatitis B and C virus, human immunodeficiency virus (HIV) and diverticulitis related parameters (C-reactive protein and procalcitonin)).
Number of new episodes of acute diverticulitis in the trial between the two MBK-01 regimens | Up to 1 year after the start of the treatment
  Diagnosis of the new episode by diagnostic imaging (computed tomography scan or ultasound) and the presence of at least one of the following symptoms: abdominal pain, vomits, intestinal obstruction, body temperature over 38ºC, constipation, elevated acute-phase reactants leukocytes higher than 11,000 cells/µL and/or C-reactive protein higher than 5mg/dl and/or procalcitonin higher than 0.2), hematochezia reported by the patient.
Occurrence of treatment-related AES between the two MBK-01 regimens during the trial | Up to 1 year after the start of the treatment
  Frequency of AES related to the treatment with MBK-01.

SECONDARY OUTCOMES:
Effect of capsule-based fecal microbiota transplantation (FMT) patient-perceived on health outcome, measured by changes in the Gastrointestinal Quality of Life Index (GIQLI) questionnaire | Day 0, 16 weeks (3 months for the MBK-01 group), 6 months and 1 year after the start of the treatment
  Changes in the GIQLI questionnaire . It consists of 36 questions with an ordinal response scale, each one from 0 to 4 (0 being the worst and 4 the best score). The questionnaire includes 5 dimensions: symptoms, physical dysfunction, emotional dysfunction, social dysfunction and treatment effects. The score for each dimension is obtained by the sum of the responses for each item, divided by the number of questions in the item. A total score, which is from 0 to 144 points, can also be obtained.
Effect of capsule-based FMT patient-perceived on health outcome, measured by changes in the SF-36 questionnaire | Day 0, 16 weeks (3 months for the MBK-01 group), 6 months and 1 year after the start of the treatment.
  Changes in the SF-36 questionnaire. It consists of 36 questions (items) divided into 8 dimensions. For each dimension (physical functioning, role limits-physical, bodily pain, general health, vitality, social functioning, role limits-emotional, mental health), the scale ranges from 0 (the worst health status for that dimension) to 100 (the best health status).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ocaña Jiménez, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain